CLINICAL TRIAL: NCT04321642
Title: The Effect of Entonox on Stages of Labor in Nulliparous Women :a Randomized Controlled Trial
Brief Title: The Effect of Entonox on Stages of Labor in Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 071
Record Dates: First submitted 2020-01-08; First posted 2020-03-25 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2019-11

CONDITIONS: ENTONOX; Nulliparous; Duration of Labor
Keywords: Entonox; Nulliiparous
MeSH Terms: interventions — Entonox

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Entonox (Experimental): Inhalation Entonox in active phase of labor ( cervical dilatation more than 5 cm ) Inhaled Entonox before true uterine contraction in 30 sec , inhaled in 4-5 times for 1 contraction
  Interventions: Drug: Entonox
- Not receive Entonox (Active Comparator): Not receive any gas when archive in active phase of labor( cervical dilatation more than 5 cm )
  Interventions: Drug: Not receive Entonox

INTERVENTIONS:
Drug: Entonox — Entonox gas with mouth piece
  Other Names: Entonox gas
  Arms: Entonox
Drug: Not receive Entonox — Not receive any gas
  Arms: Not receive Entonox

SUMMARY:
This Trial study about The effect of Entonox associated with duration of labor in Active phase and efficacy for relief pain of labor .So investigators start to study up to 14 months

DETAILED DESCRIPTION:
Investigators will enroll participants in 2 groups by randomized . First group will inhale Entonox and the second group not receive any gas . The participants in Entonox group will inhale gas in 4-5 times for each uterine contraction and Nurse will measure blood pressure , O2 saturation ,pain score before use gas . The outcome,investigators study about Apgar score , duration of labor , pain relief in both group,route of delivery and estimated blood loss

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* Age 18 years old or more
* Gestational age 37-40+6 wks
* Singleton
* Cephalic presentation
* Cervical dilatation > 5 cm
* Estimated fetal weight 2,500-4,000 gm

Exclusion Criteria:

* Estimated fetal weight more than 4,000 gm
* High risk pregnancy (Hypertension in pregnancy ,Endocrine disorder , autoimmune disorder , epilsepsy etc)
* SpO2 < 95 %
* Contraindication for Entonox usage ( Severe head injury , asthma , Pulmonary disease,Otitis media )
* Drug allergy : Metoclopramide , Dimenhydrinate , Pethidine ,Entonox

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Effect of Entonox for duration of labor | up to 14 months
  Study about duration of labor after receive Entonox in active phase of labor

SECONDARY OUTCOMES:
Rate of patients who inhaled Entonox for pain relieve | up to 14 months
  % of patients relieve pain after inhaled Entonox , Investigators measure by visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Somboon sornsukulrat, MD, Study Chair — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Entonox